CLINICAL TRIAL: NCT06650228
Title: Assessment of Knowledge of Cardiovascular Disease Risk Factors and Healthy Lifestyle Behaviours in Patients with Ankylosing Spondylitis
Brief Title: Cardiovascular Disease Risk Factors and Healthy Lifestyle Behaviours in Patients with Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-13/114
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with ankylosing spondylitis

SUMMARY:
A review of the literature did not identify any studies that assessed knowledge of cardiovascular disease risk factors and healthy lifestyle behaviours in patients with ankylosing spondylitis. The aim of this study is to assess knowledge of cardiovascular disease risk factors, healthy lifestyle behaviours and physical activity levels in patients with ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis according to ASAS diagnostic criteria
* Being aged 18-65
* Stable medication use for at least 3 months
* Voluntary participation in the study

Exclusion Criteria:

* Having uncontrolled cardiopulmonary disease
* Being pregnant
* Having undergone recent surgery
* Presence of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18-65 years who are clinically stable and diagnosed with ankylosing spondylitis according to ASAS diagnostic criteria and who are being followed up at the Rheumatology Polyclinic of the Department of Physical Medicine and Rehabilitation at Kirsehir Ahi Evran University will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge of cardiovascular disease risk factors | 10 minutes
  This will be evaluated using The Cardiovascular Disease Risk Factors Knowledge Level scale. The maximum score that can be obtained from the 28-question scale is 28.Higher scores on the scale indicate better knowledge of cardiovascular disease.
Healthy lifestyle behaviors | 15 minutes
  It will be evaluated with the Healthy Lifestyle Behaviors scale II.The lowest score on the whole scale is 52 and the highest is 208. As the score obtained from the survey increases, it is assumed that the participant's level of healthy lifestyle behaviour is high.

SECONDARY OUTCOMES:
Physical activity | 5 minutes
  Physical activity level will be evaluated using International Physical Activity Questionnaire-Short form
Cardiovascular risk | 5 minutes
  The Framingham Risk Score will be calculated to determine cardiovascular risk. Framingham risk score; if the estimated risk of cardiovascular events is above 10%, the risk is considered high; if it is below 10%, the risk is considered low.
Comorbidity | 5 minutes
  Comorbidity level will be evaluated with the Charlson Comorbidity Index

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, Principal Investigator — Kirsehir Ahi Evran University; Basak Kavalci Kol, Study Chair — Kirsehir Ahi Evran University; Figen Tuncay, Study Chair — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)